CLINICAL TRIAL: NCT01769690
Title: The Effect of Low Frequency STN DBS on Sleep and Vigilance in PD Patients
Brief Title: The Effect of Low Frequency STN DBS on Sleep and Vigilance in Parkinson's Disease (PD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Amy Amara, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: F121004006; 1K23NS080912 (NIH)
Record Dates: First submitted 2013-01-10; First posted 2013-01-17 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Parkinson's Disease
Keywords: PD; Parkinson's Disease; DBS; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant was blinded to the DBS settings during the sleep study but investigator was not; however, the investigator was blinded to the DBS setting during the interpretation of the sleep study.
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS stimulator setting alteration (Experimental)
  Interventions: Other: DBS stimulator setting alteration; Other: virtual reality simulator

INTERVENTIONS:
Other: DBS stimulator setting alteration — 2 sleep study options Phase I: Participants will undergo 2 sleep studies, one with the stimulator "on" at the subject's stable, clinically effective settings and one with the stimulator "off." the order of the "off" and "on" nights will be randomized. Although blinding will be attempted, because of the significant motor effects produced with the "on" setting, participants may be able to tell when the DBS is "OFF." In the second phase, the first sleep study night will be with the stimulator "OFF". The order of the "HIGH", and "LOW" frequency nights will be randomized 1:1 and balanced across subjects and will occur on the 2nd and 3rd PSG nights.
  Phase II Sleep study evaluation will include three nights of recording: 1) OFF with the stimulator off, 2) HIGH with the stimulator on at the participant's stable and clinically effective settings, and 3) LOW with the stimulator set at a low frequency that uses less energy
Other: virtual reality simulator — This virtual pedestrian environment is a measure of "real-world" street-crossing behavior. This simulation is composed of an elevated platform that simulates a curb at a street-side and 3 monitors (arranged in a semi-circle) on which the subject, while wearing headtracker equipment, views the virtual environment of bidirectional traffic. When the subject deems it is safe to cross the virtual street, he/she steps off the platform/curb, which activates crossing of the street by a cartoon representation of the participant. The speed of street crossing by the cartoon is determined by each individual subject's walking speed, which is measured prior to the test.
  Other Names: Wake time vigilance in PD patients

SUMMARY:
The study design is a within-subject randomized cross-over design to evaluate the effects of DBS on sleep architecture, as measured by polysomnography, and on wake-time vigilance, as measured by a virtual reality street-crossing simulator.

DETAILED DESCRIPTION:
In the proposed study, we will use a within-subject randomized clinical trial to measure objective changes in sleep architecture with DBS "on" and to compare effects of different DBS stimulation parameters on sleep architecture as measured by sleep studies. The study design will allow us to address our hypothesis that low frequency deep brain stimulation parameters are more effective than the conventional settings at improving sleep architecture and wake-time vigilance. If our hypothesis is correct, low frequency settings could be used during sleep and this would prolong stimulator battery life, therefore decreasing the frequency of required surgical battery changes for DBS. These data will be valuable in considering clinical treatment strategies and provide insight into the basic mechanisms of sleep dysfunction in PD. The study may also contribute to understanding how to achieve maximum clinical benefit from DBS while minimizing morbidity and cost.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have undergone bilateral subthalamic nucleus (STN) DBS surgery for treatment of PD.
2. Stable DBS stimulator settings and medication regimen for at least 6 weeks prior to the sleep studies.
3. Sleep dysfunction as measured by the Pittsburgh Sleep Quality Index (PSQI) (score >5)
4. 19 years of age or older
5. Ability to walk up and down stairs

Exclusion Criteria:

1. Known narcolepsy
2. Other previous surgical treatment of Parkinson's disease(with the exception of unilateral STN DBS) including pallidotomy, thalamotomy, or gene therapy procedures.
3. Pregnant women will be excluded from this study.
4. Untreated obstructive sleep apnea. If obstructive sleep apnea is discovered during the first sleep study, the subject will be removed from the study. After they have been treated for at least 6 weeks with continuous positive airway pressure (CPAP), they can re-start the study.
5. Inability to walk without assistance, including a cane, wheelchair, or walker
6. Cognitive dysfunction that would prevent subject's ability to participate in the study.
7. Blindness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Differences in sleep efficiency between the high and low frequency nights | 3 non-consecutive nights of sleep study within 4 weeks
  Phase I subjects will undergo 2 sleep studies, one with the stimulator "on" at the subject's stable, clinically effective settings and one with the stimulator "off." Phase 2 subjects will spend the first night in the sleep lab with DBS turned off. The order of the high and low frequency nights (on the second and third study nights) will be randomized.

SECONDARY OUTCOMES:
Wake-time vigilance as measured by a virtual reality street-crossing simulator | 4 weeks
  On the morning following the high and low frequency sleep study nights, subjects will evaluated with a virtual reality street-crossing simulator as a measurement of vigilance.

OTHER OUTCOMES:
Motor outcomes | 4 weeks
  Following each sleep study night, subjects will be evaluated with the Unified Parkinson's Disease Rating Scale part III at their overnight DBS settings and 30 minutes after resuming their conventional, motor effective wake-time settings.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Amara, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States